CLINICAL TRIAL: NCT05053802
Title: Efficiency and Safety of Microwave Ablation Plus Immune Checkpoint Inhibitor for Patients With Multiple Primary Lung Cancer: A Open, Multi-center, Phase II Clinical Trial
Acronym: MAGIC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Chang Chen, Shanghai Pulmonary Hospital, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L20-349
Record Dates: First submitted 2021-09-13; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Multiple Primary Lung Cancer
Keywords: MPLC; Microwave ablation; PD-1 inhibitor
MeSH Terms: interventions — camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Microwave ablation plus Camrelizumab (Experimental): Microwave ablation plus Camrelizumab (no more than 16 cycles)
  Interventions: Combination Product: Microwave ablation plus Camrelizumab
- Microwave ablation (Other): Microwave ablation
  Interventions: Device: Microwave ablation

INTERVENTIONS:
Combination Product: Microwave ablation plus Camrelizumab — Tumor received treatment of microwave ablation and received no more than 16 cycles of Camrelizumab
  Arms: Microwave ablation plus Camrelizumab
Device: Microwave ablation — Tumor received treatment of microwave ablation
  Arms: Microwave ablation

SUMMARY:
Prospective, multi-center, phase II clinical trial. The study plans to enroll 146 patients with multiple lung cancers. After signing the informed consent, they were screened to meet the admission and discharge criteria, and received microwave ablation treatment. Electromagnetic navigation bronchoscope-guided intrapulmonary microwave ablation or percutaneous microwave ablation was selected according to the patient's wishes and the evaluation of the surgeon. After the operation, they were randomized and the experimental group accepted PD-1 immune checkpoint inhibitor treatment (microwave ablation combined with Camrelizumab treatment does not exceed 16 cycles, or disease progression/worsening or confirmed imaging disease progression, or withdrawal for any reason), the control group does not After receiving any treatment, the two groups were followed up closely (36 months after the last treatment, including safety follow-up and survival follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. 18～79 years old;
2. Multiple pulmonary nodules diagnosed by CT, the number of target lesions ≥2 and ≤5 (definition of target lesions: the largest diameter of a single nodule ≥8 mm or the largest diameter of a solid component ≥5mm, and the largest single nodule Diameter ≤30 mm), the target lesions are distributed in at least two lung lobes;
3. The target lesions need to be pathologically indicated as lung cancer, and at least one of the target lesions is pathologically diagnosed as lung cancer (at least one target lesion is pathologically diagnosed as lung cancer, and the CT follow-up after anti-inflammatory treatment for the remaining target lesions is clear and stable for no less than 3 months, which is also consistent with the entry Group conditions);
4. The patient has no lymph node metastasis, lung metastasis or distant organ metastasis (N0, M0);
5. ECOG PS score 0-2;
6. Expected survival time ≥ 12 months;
7. Sufficient hematology function, defined as absolute neutrophil count ≥1.5×109/L, platelet count ≥80×109/L, hemoglobin ≥90g/L (no history of blood transfusion within 7 days, no G-CSF and others Correction of hematopoietic stimulating factors);
8. Sufficient liver function, defined as all patients with total bilirubin level ≤1.5 times upper limit of normal (ULN) and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤2.5 times ULN;
9. Sufficient renal function, defined as creatinine clearance ≥50ml/min (Cockcroft-Gault formula);
10. The coagulation function is adequate, defined as the international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN; if the subject is receiving anticoagulation therapy, as long as the INR/PT is within the proposed range of anticoagulation drugs Can;
11. For female subjects of childbearing age, the urine or serum pregnancy test should be negative within 3 days before receiving the first study drug administration. If the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is required;
12. If there is a risk of conception, male and female patients need to use high-efficiency contraception (that is, a method with a failure rate of less than 1% per year) and continue until at least 180 days after stopping the trial treatment;
13. Subjects voluntarily join the study and sign written informed consent before any trial-related procedures are implemented. They have good compliance and cooperate with follow-up.

Exclusion Criteria:

1. Genetic testing is positive for at least one mutation of EGFR, ALK, ROS1 fusion, BRAF V600E mutation, and NTRK fusion;
2. Pulmonary nodules with the largest diameter> 30mm in preoperative imaging examination;
3. Preoperative imaging examination or mediastinal lymph node puncture indicates patients with positive preoperative lymph nodes;
4. Patients with distant metastasis or chest or ascites found in preoperative examination;
5. Currently participating in interventional clinical research treatment, or receiving treatment with other research drugs or research devices within 3 months before the first intervention;
6. Any systemic anti-tumor treatment before tumor ablation, including interventional chemoembolization, radiotherapy, chemotherapy, targeted therapy, or Chinese patent medicine with anti-tumor indications or immunomodulatory drugs (thymosin, interferon, interleukin, etc.) ), or received major surgery within 3 weeks before the first intervention;
7. Have received the following therapies in the past: anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or drugs that stimulate or synergistically inhibit T cell receptors (for example, CTLA4, OX-40, CD137);
8. There are multiple factors that affect surgery or ablation (such as coagulation dysfunction, immune system disease, etc.);
9. Abnormal coagulation function (PT>16 s, APTT>43 s, TT>21 s, Fbg< 2 g/L), bleeding tendency (such as active peptic ulcer) or receiving thrombolytic or anticoagulant therapy;
10. Pulmonary hemorrhage ≥ CTCAE grade 2 occurred within 4 weeks before the first intervention; other parts of hemorrhage ≥ CTCAE grade 3 occurred within 4 weeks before treatment;
11. Known history of human immunodeficiency virus (HIV) infection (ie HIV 1/2 antibody positive), known syphilis infection (syphilis antibody positive), active tuberculosis, active hepatitis without treatment;
12. People with severe impairment of heart, liver, and kidney functions (heart function grades 3 to 4, ALT and/or AST are more than 3 times the upper limit of normal, and Cr exceeds the upper limit of normal);
13. Known mental illness or drug abuse that may affect compliance with test requirements;
14. Patients with other malignant tumors or hematological diseases;
15. Pregnant, planned pregnancy and breast-feeding female patients (when urine HCG>2500IU/L, it is diagnosed as early pregnancy);
16. The investigator believes that it is not suitable for inclusion.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2021-03-21 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
1 Year Recurrence-free survival | 1 year
3 Year Recurrence-free survival | 3 years
Progression-free rate of remaining lesions | 5 years

SECONDARY OUTCOMES:
2 Year Recurrence-free survival | 2 years
5 Year Recurrence-free survival | 5 years
3 year overall survival | 3 years
5 year overall survival | 5 years
Complication rate | 3 years
Quality of life score | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Chang Chen, Dr, Study Chair — Shanghai Pulmonary Hospital, Shanghai, China
Locations (6):
- China (6):
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai, Shangh

IPD SHARING:
Plan to Share IPD: Undecided